CLINICAL TRIAL: NCT06851247
Title: Toripalimab Plus Anlotinib Combined with GP Induction Chemotherapy and Concurrent Chemoradiotherapy Followed by Toripalimab Maintenance Therapy for High-risk, Locally Advanced Nasopharyngeal Carcinoma：A Single-arm, Phase II Clinical Trial
Brief Title: GAPP Induction and Concurrent Chemoradiotherapy Followed by Toripalimab Maintenance for Nasopharyngeal Carcinoma.
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, YiJun Hua, Chief Physician, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-FXY-171-NPC
Record Dates: First submitted 2025-02-23; First posted 2025-02-28 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — toripalimab; anlotinib; Gemcitabine; Cisplatin; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental group (Experimental): Toripalimab Plus Anlotinib Combined With GP Induction Chemotherapy and Concurrent Chemoradiotherapy Followed by Toripalimab Maintenance Therapy
  Interventions: Drug: Toripalimab; Drug: Anlotinib; Drug: Gemcitabine; Drug: Cisplatin; Radiation: radiation

INTERVENTIONS:
Drug: Toripalimab — Fixed dose: 240mg/ time, add 100ml normal saline, intravenous infusion for 30 minutes (not less than 20 minutes, not more than 60 minutes).
  The first course of induction chemotherapy (D1) is used on the first day of each cycle, and every 21 days is a course of treatment up to 18 courses or one year.
  After intravenous infusion of triplelizumab, GP regimen induction chemotherapy was administered at an interval of 30-60 minutes.
Drug: Anlotinib — Oral administration before breakfast, 10mg/ time/day, once a day (d1-14), repeated every 3 weeks, using three courses, one week before radiotherapy discontinuation.
  Use on the day the first course of induction chemotherapy begins (D1).
Drug: Gemcitabine — 1000mg/m2, D1, D8, add 0.9% normal saline 500ml, intravenous infusion. Every 21 days is a treatment cycle. If the recovery of toxicity in the subject is not sufficient for the next course of chemotherapy, the start of the next course of chemotherapy may be appropriately delayed, but the delay cannot exceed 21 days.
  The treatment was continued for 3 courses.
Drug: Cisplatin — Induction Chemotherapy: 80mg/m2, D1, add 1000ml 0.9% normal saline, intravenous infusion for 3 hours.
  Concurrent Chemoradiotherapy100mg/m2, add 5% glucose 500ml, intravenous drip. Use on the first day of each cycle, every 21 days for a treatment cycle
Radiation: radiation — IMRT, 33Fx

SUMMARY:
In order to explore the efficacy and safety of targeted therapy and immunotherapy combined with GP chemotherapy in the treatment of high risk advanced nasopharyngeal carcinoma, the investigators design a single-arm, Phase II clinical trial targeted high-risk patients with local stage nasopharyngeal carcinoma (stage IVa: TanyN3M0/T4N0-2M0,8th AJCC/UICC staging) for Toripalimab Plus Anlotinib Combined With GP Induction Chemotherapy and Concurrent Chemoradiotherapy Followed by Toripalimab Maintenance Therapy.

DETAILED DESCRIPTION:
In order to explore the efficacy and safety of targeted therapy and immunotherapy combined with GP chemotherapy in the treatment of high risk advanced nasopharyngeal carcinoma, the investigators design a single-arm, Phase II clinical trial targeted high-risk patients with local stage nasopharyngeal carcinoma (stage IVa: TanyN3M0/T4N0-2M0,8th AJCC/UICC staging) for Toripalimab Plus Anlotinib Combined With GP Induction Chemotherapy and Concurrent Chemoradiotherapy Followed by Toripalimab Maintenance Therapy. The investigators focus on the 2-year PFS as the primary outcome.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily participate in and sign informed consent in person.
* Age 18-65, male or non-pregnant female.
* Pathological diagnosis of nasopharyngeal non-keratonic carcinoma (differentiated or undifferentiated, i.e., WHO type II or III).
* First treatment patients who did not receive antitumor therapy had no history of other malignant tumors;
* Stage IVa: TanyN3M0/T4N0-2M0 (8th AJCC/UICC stage)
* ECOG score 0-1, no serious dysfunction of heart, lung, liver, kidney and other vital organs.
* Hemoglobin (HGB) ≥90 g/L, white blood cells (WBC) ≥4.0×109 /L, platelets (PLT) ≥100×109 /L.
* Liver function: ALT and AST< 2.5 times the upper limit of normal (ULN), total bilirubin <2.0×ULN.
* Renal function: serum creatinine <1.5×ULN.

Exclusion Criteria:

* Patients with recurrent and distant metastasis of nasopharyngeal carcinoma.
* The pathology was keratinized squamous cell carcinoma (WHO type I).
* Received systemic or local glucocorticoid therapy within 4 weeks prior to enrollment.
* Participants who had participated in other drug clinical trials within 3 months before treatment.
* Patients with a known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation;
* Patients with idiopathic pulmonary fibrosis, drug-induced pneumonia, institutional pneumonia (i.e., bronchiolitis obliterans), radiation pneumonia with clinical symptoms or requiring steroid treatment, active pneumonia, or other moderate to severe lung diseases that seriously affect lung function
* Have a comorbiditis that requires long-term treatment with immunosuppressive drugs or systemic or local use of immunosuppressive doses of corticosteroids.
* Prior use of anti-PD-1 antibodies, anti-PD-L1 antibodies, anti-PD-L2 antibodies, or anti-CTLA-4 antibodies (or any other antibody that acts on the T-cell co-stimulation or checkpoint pathway), and efficacy was assessed as progressive at enrollment.
* The subject has any active autoimmune disease or history of autoimmune disease (including but not limited to: interstitial pneumonia, uveitis, enteritis, hepatitis, hypophysitis, nephritis, hyperthyroidism, hypothyroidism; Patients with vitiligo or who had complete remission of asthma in childhood and did not require any intervention as adults were included; Patients with asthma requiring medical intervention with bronchodilators were not included).
* Positive HBV DNA copy number was detected in HIV-positive patients and HBsAg positive patients (quantitative detection ≥ 1000cps/ml); Chronic hepatitis C blood screening positive (HCV antibody positive) with HCV RNA positive detection.
* Received any anti-infection vaccine (such as influenza vaccine, chickenpox vaccine, etc.) within 4 weeks before enrollment.
* Pregnancy test positive women of childbearing age and breastfeeding women.
* Patients who are unable to cooperate with regular follow-up due to psychological, social, family and geographical reasons.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Estimated)
Dates: Start 2025-01-03 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
2-year progression-free survival | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 2 years.
  2-year progression-free survival

CONTACTS AND LOCATIONS:
Locations (1):
- Sun yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
Researchers who has been approved can share